CLINICAL TRIAL: NCT04050033
Title: Clinical Study to Evaluate the Performance of Evoke Radiofrequency Device for Improvement of Skin Appearance
Brief Title: Evoke Radiofrequency Device for Improvement of Skin Appearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO608679A
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Improvement of Skin Appearance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Enrolled subjects will undergo up to 3 successive bi-weekly (every 2 weeks) treatments (Tx.1, Tx.2 and Tx.3).
  Interventions: Device: Evoke Device

INTERVENTIONS:
Device: Evoke Device — Subjects will undergo treatment with Evoke Device

SUMMARY:
The aim of the study is to evaluate the safety, efficacy, patient comfort and patient satisfaction after Evoke treatment

ELIGIBILITY:
Inclusion Criteria:

* - Signed informed consent to participate in the study.
* Female and male subjects, 35 - 75 years of age at the time of enrolment
* If female, not pregnant, lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
* In addition, negative urine pregnancy test as tested before each treatment and at the last visit for women with childbearing potential (e.g. not menopause).
* General good health confirmed by medical history and skin examination of the treated area.
* Willing to have photographs and images taken of the treated areas to be used de-identified in evaluations, publications and presentations.
* The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other aesthetic treatment methods for the last 6 months and during the entire study period.

Exclusion Criteria:

* - Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* Permanent implant in the treated area such as metal plates and screws, silicone implants or an injected chemical substance, unless deep enough in the periostal plane.
* Current or history of skin cancer, or current condition of any other type of cancer, or premalignant moles.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy and nursing.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies or use of anticoagulants in the last 10 days.
* Any surgery in treated area within 3 months prior to treatment.
* Six months delay is required if other recent treatments like light, CO2 laser or RF were performed on the same area.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with Change in Skin Appearance | 1 month, 3 month, 6 months
  Picture evaluation by blinded investigators.
Evaluate rate of Change in Skin Appearance using 3D Photographic analysis | 1 month, 3 month, 6 months
  3D Photographic analysis will be conducted using QuantifiCare System
Evaluate changes in skin using VivoSight Optical Coherence Tomography (OCT) software | 1 month, 3 month, 6 months
  Non-invasive in vivo skin imaging will be taken with the VivoSight Optical Coherence Tomography (OCT).
Evaluate changes in skin appearance comparing photographs using Mechanical Turk (MTurk). The pictures will be sent through the system and evaluated by crowd workers. | 1 month, 3 month, 6 months
  The pictures will be sent through the system and evaluated by crowd workers.

SECONDARY OUTCOMES:
Evaluate Investigator assessment of the skin appearance improvement | 1 Month, 3 Months, 6 Months
  Investigator assessment of the skin appearance improvement comparing pre and post treatment using 0 - 4 -points Likert scale at 1 month, 3 months and 6 months follow up visits:
  • 4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement; 0 = No difference
Evaluate Subject assessment of improvement and satisfaction | 1 Month, 3 Months, 6 Months
  Improvement assessment will be performed independently by the subject himself 4 points Likert scale questionnaire (Global Aesthetic Improvement Scale), as follows:
  • 4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement; 0 = No difference.
  Subject assessment of satisfaction will be filled out by subjects using a 5-points Likert scale, as follows:
  • +2 = Very satisfied; +1 = Satisfied; 0 = Indifferent; -1 = Disappointed; -2 = Very disappointed.
Evaluate histological changes to treatment area skin | 3 Months
  Positive changes in histologic evaluation: up to 5 subjects will undergo biopsies of the treated area for histology at baseline and at 3M follow-up visit. Histological sections will be stained using elastin, H&E and other collagen specific stains.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Dayan, MD, Principal Investigator — Avance Plastic Surgery Institute 5570 Longley Lane, Suite A Reno, NV 89511; Christopher Chia, MD, Principal Investigator — BodySculpt 128 Central Park S New York, NY 10019
Locations (3):
- United States (3):
  - Avance Plastic Surgery Institute, Reno, Nevada
  - Union Square Laser Dermatology, New York, New York
  - BodySculpt, New York, New York